CLINICAL TRIAL: NCT06031649
Title: Lumbar Paraspinal Muscular Properties After Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Lecturer of Physical Therapy for Women's Health, South Valley University
Other Study IDs: Lumbar Paraspinal Muscles
Record Dates: First submitted 2023-08-25; First posted 2023-09-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: 30 mother underwent cesarean section
  Interventions: Device: MyotonPRO device
- Group B: 30 healthy females who were in the control group
  Interventions: Device: MyotonPRO device

INTERVENTIONS:
Device: MyotonPRO device — It is a valid and reliable device for measuring the muscular mechanical properties
  Other Names: Myotonometry

SUMMARY:
The biomechanical characteristics of lumbar paraspinal muscles may give us insight into different lower back dysfunctions in postpartum mothers after cesarean section.

DETAILED DESCRIPTION:
Stiffness and elasticity are two mechanical characteristics of the muscles, whereas relaxation time and creeping are two viscoelastic characteristics.

Different studies investigated the mechanical properties of lumbar paraspinal muscles in numerous musculoskeletal conditions, however, no previous studies investigated these characteristics after cesarean section, which is associated with high prevalence of lower back pain when compared with normal delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women who experienced cesarean section at least for one time
* Women Who are free of specific lower back disorders
* Women who are below 34 years old and above 20 years old

Exclusion Criteria:

* Women who experienced normal vaginal birth
* Women who complain of a specific lower back disorder
* Women who are above 34 years old or below 20 years old
* Women who have a body mass index above 30 Kg/m2

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — A study in the scope of physiotherapy for women's health
Study Population: 60 females participated in this research, aged between 20 and 34 years old. They were free of specific lower back disorders. They were recruited from the outpatient clinics of South Valley Hospitals
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Lumbar Paraspinal Muscles Stiffness, measured by the MyotonPRO device in units of N/m. | 6-12 weeks after cesarean section
  muscular stiffness refers to muscle resistance against forces that deform it.
Lumbar Paraspinal Muscles Elasticity, measured by the MyotonPRO device in a relative unit | 6-12 weeks after cesarean section
  Muscular Elasticity refers to the muscular ability to return to its original shape after the removal of tensional forces.

SECONDARY OUTCOMES:
Lumbar Paraspinal Muscles Stress Relaxation Time, measured by the MyotonPRO device in milliseconds | 6-12 weeks after cesarean section
  relaxation time is a viscoelastic characteristic of the muscles, it refers to the time taken to return to the original shape after the removal of the deformative forces.
Lumbar Paraspinal Muscles Creep, measured by the MyotonPRO device in a relative unit | 6-12 weeks after cesarean section
  Muscular creep refers to the muscular ability to lengthen when constant stresses applied to it.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Deun B, Hobbelen JSM, Cagnie B, Van Eetvelde B, Van Den Noortgate N, Cambier D. Reproducible Measurements of Muscle Characteristics Using the MyotonPRO Device: Comparison Between Individuals With and Without Paratonia. J Geriatr Phys Ther. 2018 Oct/Dec;41(4):194-203. doi: 10.1519/JPT.0000000000000119. PMID 28005829
- [Background] Struzik A, Karamanidis K, Lorimer A, Keogh JWL, Gajewski J. Application of Leg, Vertical, and Joint Stiffness in Running Performance: A Literature Overview. Appl Bionics Biomech. 2021 Oct 21;2021:9914278. doi: 10.1155/2021/9914278. eCollection 2021. PMID 34721664
- [Background] Parikh S, Suchi J. Prevalence of low back pain and its impact on quality of life in post-partum women. International Journal of Scientific Research. 2016; 7:14342-8.